CLINICAL TRIAL: NCT05481151
Title: A Phase IIIb, Randomized, Open-Label, Parallel Group, Multicenter Study to Assess Efficacy, Safety, and Tolerability of Two Dosing Regimens of Ropeginterferon Alfa-2b-njft (P1101) in Adult Patients With Polycythemia Vera (PV)
Brief Title: A Study to Assess Efficacy, Safety, and Tolerability of P1101 in Adult Patients With PV
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECLIPSE PV / A22-203
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Polycythemia Vera
Keywords: Polycythemia Vera; Essential Thrombocythemia; P1101; Ropeginterferonalfa-2b-njft; Polycythemia; Vera; PharmaEssentia; Besremi; Ropeg
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Polycythemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- P1101 250-350-500mcg (Experimental): Pre-filled Syringe, Q2W starting at 250-350-500, SC injection
  Interventions: Drug: P1101 (Ropeginterferon alfa-2b-njft)
- Ropeginterferon alfa-2b-njft (Active Comparator): Pre-filled Syringe, Q2W starting at 100 up to 500 (50mcg increases), SC injection
  Interventions: Drug: Ropeginterferon alfa-2b-njft (P1101)

INTERVENTIONS:
Drug: P1101 (Ropeginterferon alfa-2b-njft) — Ropeginterferon alfa-2b-njft
  Arms: P1101 250-350-500mcg
Drug: Ropeginterferon alfa-2b-njft (P1101) — Ropeginterferon alfa-2b-njft
  Arms: Ropeginterferon alfa-2b-njft

SUMMARY:
A Study to Assess Efficacy, Safety, and Tolerability of P1101 in Adult Patients with PV

DETAILED DESCRIPTION:
Polycythemia vera (PV) is the most common type of chronic myeloproliferative neoplasm (MPN), with an annual reported incidence of up to 2.6/100,000. This is a long-term debilitating and life-threatening disease because it is associated with the risk of thrombosis, bleeding, and progression to myelofibrosis (MF) and secondary acute myeloid leukemia (sAML)

Ropeginterferon alfa-2b-njft (P1101), which gained US marketing authorization in November 2021, is the only interferon alfa approved for the treatment of PV.

This study aims to evaluate the efficacy, tolerability, and safety of ropeginterferon alfa-2b-njft (P1101) in US and Canadian PV patients, utilizing an optimized dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18 years at the time of signing the informed consent form
2. Subjects diagnosed with PV according to the 2008 or 2016 World Health Organization (WHO) criteria
3. Subjects with good liver function at screening, which is defined as total bilirubin ≤1.5 × upper limit of normal (ULN), international normalized ratio (INR) ≤1.5 × ULN, albumin >3.5 g/dL, alanine aminotransferase (ALT) ≤2.0 × ULN, and aspartate aminotransferase (AST) ≤2.0 × ULN
4. Hemoglobin (HGB) ≥10 g/dL for females, and HGB ≥11 g/dL for males at screening
5. Neutrophil count ≥1.5 × 10^9/L at screening
6. Creatinine clearance rate ≥40 mL/min at screening (according to the Cockcroft-Gault formula)
7. Males and females of childbearing potential, as well as all women <2 years after the onset of menopause, must agree to use an acceptable form of birth control until 60 days following the last dose of the study drug, and females must agree to not breastfeed during the study
8. Written informed consent obtained from the subject and ability for the subject to comply with the requirements of the study

Exclusion Criteria:

1. Any contraindications to interferon alfa or hypersensitivity to interferon alfa
2. Subjects who stopped prior to interferon alfa therapy due to low efficacy or poor tolerability
3. Subjects with severe or serious diseases that the Investigator determines may affect the subject's participation in this study
4. History of major organ transplantation
5. Pregnant or breastfeeding women
6. Subjects with any other diseases that the Investigator determines will affect the study results or may weaken the compliance to protocol, including but not limited to:

   1. Prior or current autoimmune thyroid disease (clinical symptoms of hyper- or hypo-thyroidism), except subjects with controlled thyroid replacement therapy, could be enrolled
   2. Other documented autoimmune diseases (such as hepatitis, immune thrombocytopenia [ITP], scleroderma, psoriasis, or any autoimmune arthritis)
   3. Clinically significant pulmonary infiltration, infectious pneumonia, and non-infectious pneumonia, or a past history of interstitial pneumonia at screening
   4. Active infection with systemic manifestations (e.g., presence of bacteria, fungi, and/or human immunodeficiency virus [HIV] at screening, excluding hepatitis B [HBV] and/or hepatitis C [HCV] at screening)
   5. Evidence of severe retinopathy (e.g., cytomegalovirus [CMV]-induced retinitis, macular degeneration) or clinically significant eye diseases (due to diabetes or hypertension)
   6. History or presence of clinically relevant depression per Investigator's judgment
   7. Previously had suicidal attempts or has any risk for suicidal tendency at screening
   8. Poorly controlled diabetes defined as HbA1c >8.0% for at least 1 year
   9. Active thromboembolic complications caused by PV and abdominal hemorrhage in the active phase
   10. History of any malignancy within 5 years (except adequately treated non-melanoma skin cancer, prostate cancer status post resection with an undetectable prostate-specific antigen (PSA), curative treated in-situ cancer of the cervix, ductal carcinoma in situ (DCIS) of the breast, Stage 1 Grade 1 endometrial carcinoma, or other solid tumors including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥2 years prior to study)
   11. History of alcohol or drug abuse in the past year
   12. History or evidence of post-polycythemia vera-myelofibrosis (PPV-MF), essential thrombocythemia, or any non-PV MPN
   13. Presence of blast cells in the peripheral blood in the past 12 weeks
7. Use any investigational drug <4 weeks prior to the first dose of study drug, or not recovered from effects of prior administration of any investigational drug
8. Any subject requiring a legally authorized representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Compare efficacy, safety, and tolerability of P1101 utilizing 250-350-500 mcg compared to the current labeled dosing through assessing the proportion of subjects that are in a complete hematologic response at Week 24. | 24 weeks
  CHR is defined as hematocrit (HCT) <45%, white blood cell (WBC) count <10 × 10^9/L, platelets (PLT) ≤400 × 10^9/L in the absence of phlebotomy in the previous 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Ole Zagrijtschuk, MD, PhD, Study Director — PharmaEssentia Corporation
Locations (23):
- United States (17):
  - Baptist MD Anderson, Jacksonville, Florida
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - University of Kansas Medical Center, Westwood, Kansas
  - Mercy Health, Paducah, Kentucky
  - Tulane University Medical Center, New Orleans, Louisiana
  - American Oncology Partners of Maryland PA (Center for Cancer & Blood Disorders), Bethesda, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Astera HealthCare, East Brunswick, New Jersey
  - Mount Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest Baptist Medical Center, High Point, North Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - MD Anderson, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia - Emily Couric Cancer Center, Charlottesville, Virginia
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Juravinski Cancer Center - Hamilton Health Sciences, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No